CLINICAL TRIAL: NCT06103968
Title: Determining the Influence Gastric Tube Presence in Upholding the Correct Placement of LMA Blockbuster During Surgery.
Brief Title: Influence of Gastric Tube Presence in Upholding the Correct Placement of LMA Blockbuster
Status: Completed | Type: Observational
Sponsor: Aligarh Muslim University (Other)
Responsible Party: Principal Investigator, MUAZZAM HASAN, Assitant Professor, Aligarh Muslim University
Other Study IDs: LMA Blockbuster
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LMA BLOCKBUSTER — In this study we wish to evaluate weather gastric tube inserted through LMA helps in maintaining the LMA blockbuster placement by comparing fibreoptic bronchoscope (FOB) scores recorded immediately after LMA placement and at the end of the surgical procedure.
  Other Names: GASTRIC TUBE

SUMMARY:
Since its invention in 1981 by Dr. Archie Brain, the classical laryngeal mask airway (LMA ) has undergone many modifications. Today various LMAs are available that can also help in Ryle's tube insertion, intubation via LMA, deep extubation, adjunct in difficult airway and for spontaneous ventilation in short procedures.

One of the newer modifications is the Blockbuster LMA. It was invented by Prof. Ming Tian, the president of Chinese Difficult Airway Society and is being increasingly used for cases of difficult intubation. It has some unique features like its 95 degrees angulated airway that makes it easier to insert. It also has a gastric port and provides better sealing pressures at lower volumes.

However the one of the major concern with supraglottic airway is that despite correct placement it may dislodge, or its position may change intraoperatively especially in surgeries where patient position needs to be changed or patient is moved/transferred or head and neck surgeries.

In this study investigator wishes to evaluate weather gastric tube inserted through LMA helps in maintaining the LMA blockbuster placement by comparing fibreoptic bronchoscope (FOB) scores recorded immediately after LMA placement and at the end of the surgical procedure.

DETAILED DESCRIPTION:
Following approval by the Board of studies, Department of anaesthesiology and ethical committee of this institution the study will be conducted in J N Medical College and hospital on 60 patients undergoing operative procedures under general anaesthesia. Patients will be included in the study after well informed written consent, including the information that they would be part of this ongoing institutional research.

STUDY DESIGN Prospective randomised controlled study

STUDY POPULATION The study will be conducted on 60 patients admitted to JNMCH, AMU Aligarh planned for operative procedure under general anaesthesia.

In this study investigator wishes to evaluate weather gastric tube inserted through LMA helps in maintaining the LMA blockbuster placement by comparing fibreoptic bronchoscope (FOB) scores recorded immediately after LMA placement and at the end of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA Grade I & II patients
* Age between 20-70 years
* Weight between 40-70 kg
* Patients of both sexes
* All classes of MP Grades

Exclusion Criteria:

* Any pathology of the oral cavity that may obstruct the insertion of device
* Mouth opening less than 2.5cm.
* Potentially full stomach patients (trauma, morbid obesity, history of gastric regurgitation and heart burn, full term pregnancy)
* risk of oesophageal reflux (hiatus hernia)
* Bleeding disorder
* Unable to provide informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 60 patients admitted to JNMCH, AMU Aligarh planned for operative procedure under general anaesthesia.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
POGO SCORE | IMMEDIATELY AFTER LMA PLACEMENT AND AT THE END OF SURGERY JUST BEFORE REMOVAL OF LMA
  Grading the placement of LMA blockbuster through Fibreoptic Bronchoscope score of at the start and end of the surgery.

SECONDARY OUTCOMES:
GASTRIC TUBE INSERTION SUCCESS RATE | within 2 minutes of LMA Blockbuster placement
  Ease and success rate of gastric tube insertion; number of attempts taken if successfull

CONTACTS AND LOCATIONS:
Overall Officials: MUAZZAM HASAN, MD, Principal Investigator — AMU
Locations (1):
- Jawaharlal Nehru Medical College, Aligarh, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Patient particulars, PAC sheets and informed consent.

REFERENCES:
- [Result] Brimacombe J, Vosoba Judd D, Tortely K, Barron E, Branagan H. Gastric tube-guided reinsertion of the ProSeal laryngeal mask airway. Anesth Analg. 2002 Jun;94(6):1670. doi: 10.1097/00000539-200206000-00062. No abstract available. PMID 12032052